CLINICAL TRIAL: NCT01070602
Title: The Effect of Anterior Corneal Incisions on Intraoperative Floppy Iris Syndrome (IFIS) Incidence and Severity in Tamsulosin Treated Cataract Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRIFIS-001
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-03

CONDITIONS: Intraoperative Floppy Iris Syndrome
Keywords: IFIS

ARMS (1):
- anterior corneal incision (Experimental)
  Interventions: Procedure: anterior (more central) corneal paracentesis incision

INTERVENTIONS:
Procedure: anterior (more central) corneal paracentesis incision — 3 corneal paracentesis incisions will be located 1 mm anterior to the limbus.

SUMMARY:
Intraoperative Floppy Iris Syndrome (IFIS) may occur during cataract surgeries in patients treated with alpha 1 blockers. IFIS related to alpha 1 blocker Tamsulosin (used for prostate hypertrophy) was reported in 50-90% of patients. IFIS during surgery make the surgery more difficult and raise complication rate.

Using anterior corneal incisions was reported briefly in literature as a prophylactic means but was not studied prospectively. we believe (according to our clinical experience) that these anterior incisions do help to reduce the incidence and severity of IFIS signs and complications rate during surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. cataract candidates treated (in the present or in the past) with tamsulosin
2. aged 55 or more
3. candidates for topical anesthesia
4. no allergy to anticholinergic or adrenergic drugs
5. able to understand and sign an informed consent

Exclusion Criteria:

1. history of uveitis
2. iris neovascularization
3. s/p iris surgery
4. traumatic/uveitis induced cataract
5. dialysis / abscence of zonules

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
the number of IFIS cases observed during operation. | during the operations

SECONDARY OUTCOMES:
assessing the clinical grade of observed IFIS cases | during the operations

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel